CLINICAL TRIAL: NCT06131515
Title: Efficacy of Extracorporeal Shock Wave Therapy on Carpal Tunnel Syndrome Post Mastectomy Lymphedema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shahira Sami, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1582017
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (experimental group) (Experimental): This group includes 34female patients who will receive extra corporeal shock wave therapy one session per week for 4 weeks in addition to physical therapy exercises (including carpal bone mobilization, nerve glide skin care and manual lymph drainage 2 sessions per week for 4 weeks.
  Interventions: Device: extra corporeal shock wave therapy device
- Group B (control group) (Experimental): This group includes 34female patients who will receive shame extra corporeal shock wave therapy one session per week for 4 weeks in addition to physical therapy exercises (including carpal bone mobilization, nerve glide exercises, skin care and manual lymph drainage 2 sessions per week for 4 weeks.
  Interventions: Device: extra corporeal shock wave therapy device

INTERVENTIONS:
Device: extra corporeal shock wave therapy device — Patients were seated in a relaxed position with their forearm and finger placed on the table. The median nerve was identified at the pisiform level of the proximal carpal tunnel, with the palm facing upwards. rESWT was delivered with the Physio Shock Wave Therapy system .The rESWT probe was located and oriented perpendicularly on the median nerve, and treatment comprised graduated shots at a bar pressure of 4 and a pulse repetition frequency of 5Hz for each patient ( The treated area was parallel to the median nerve from the pisiform level to 2 cm proximal to the inlet of the carpal tunnel with equal diffusion of 800, 900, 1000, 1100 shots from first to fourth session respectively. The procedure was painless, and there was no need for additional anesthesia or analgesia.
  In the control group, sham rESWT just made the same sound without energy emission

SUMMARY:
Sixty eight female patients who had symptoms of carpal tunnel syndromesuch as wrist pain or numbness and paraesthesia and had lymphedema of an upper extremity.Their ages will be ranged from 40 to 60 years. The participants will be selected from Out Patient clinic of Faculty of Physical Therapy, Cairo University and randomly distributed into two equal groups.Duration of treatment for 4weeks.All subjects signed an informed consent form, and the rights of subjects were protected.

DETAILED DESCRIPTION:
In this study the patients will be randomly assigned into two equal groups(34 patients for each group)Group A (experimental group):This group includes 34female patients who will receive extra corporeal shock wave therapy one session per week for 4 weeks in addition to physical therapy exercises (including carpal bone mobilization, nerve glide skin care and manual lymph drainage 2 sessions per week for 4 weeks. Group B (control group):

This group includes 34female patients who will receive shame extra corporeal shock wave therapy one session per week for 4 weeks in addition to physical therapy exercises (including carpal bone mobilization, nerve glide exercises, skin care and manual lymph drainage 2 sessions per week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

All participants could be considered and enrolled if they conformed to the diagnosis of CTS, with clinical symptoms for at least 3 months.

The clinical symptoms and signs for the diagnosis of CTS were as follows:

1. Paresthesias and painful swelling with weakness of the affected hand, exacerbated while sleeping or by repetitive use of the wrist, which would be relieved by shaking the hand with postural change.
2. Sensory loss with numbness in the regions of the hand innervated by the median nerve;
3. Impaired motor function with atrophy of the median nerve-innervated thenar muscles.
4. Positive Tinel's sign.

The subject selection will be according to the following criteria:

* Female patient their age range between 40-60 years.
* Symptoms of CTS as pain, tingling sensation for at least 3 months.
* Unilateral or bilateral Lymphedema following mastectomy
* All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

* The potential participants will be excluded if they meet one of the following criteria:
* Local infections at the hand level.
* Patients with prior medical histories of cardiac arrhythmias.
* Patient with venous thrombosis.
* Areas of skin with lesions and impaired sensation
* Other diseases that cause significant swelling.
* During pregnancy and breastfeeding.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Nerve conduction studies | 4weeks
  For assessing the motor response, the recorder electrode on abductor pollicis brevis muscle and median nerve was stimulated at wrist region with stimulator electrode, 8 cm proximal to the active electrode , and the distal latency was recorded. Regarding the sensory response, the recorder was fastened on the third finger, and stimulator electrode was placed 14 cm proximal to the recorder and stimulated median nerve at wrist and at palm region, then distal latency was recorded. If only the SNAP distal latency was long, patient had mild CTS, but if both SNAP and CMAP distal latency were long and denervation was not observed in electromyography of APB, it was moderate CTS
Limb volume | 4weeks
  Upper limb volumes were calculated from circumference measurements taken at 5cm intervals from the dorsum of the wrist to the axilla. Volume was calculated from circumference using the established formula
Visual analogue scale (VAS) | 4weeks
  The VAS uses a straight 10-centimeter line with one end being 'no pain' and on the other end the 'worst imaginable pain'. The patient chooses a spot on the line then places a perpendicular line to indicate their pain level within the last 24 hours.
Boston Carpal Tunnel Questionnaire (BCTQ) | 4weeks
  The BCTQ is used to evaluate symptom severity and dysfunction in patients with CTS .It contains 2 measurement scales: a symptom severity scale (BCTQ-S) and a functional status scale (BCTQ-F). The BCTQ-S uses 11 questions to evaluate the intensity and frequency of pain, numbness, weakness and loss of dexterity on a five-point scale ranging from 1 (no symptoms) to 5 (severe symptoms). The results are interpreted as the average scores of the 11 questions. The BCTQ-F has 8 questions to evaluate the level of difficulty in performing daily tasks, each rated on a five-point scale ranging from 1 (no difficulty) to 5 (cannot do at all due to hand or wrist symptoms). The results are interpreted as the average scores of the 8 questions

CONTACTS AND LOCATIONS:
Overall Officials: shahira sami, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Khadra Mohamed Ali, Cairo
  - Shahira Sami, Cairo

IPD SHARING:
Plan to Share IPD: Yes
after 6months we will share the study protocol and informed consent.
Supporting Information: Study Protocol, ICF
Time Frame: after 6 months of study